CLINICAL TRIAL: NCT00095225
Title: A Phase II, Multicenter, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Bevacizumab in Combination With Chemotherapy (Docetaxel or Pemetrexed) or Tarceva (Erlotinib) Compared With Chemotherapy (Docetaxel or Pemetrexed) Alone for Treatment of Recurrent or Refractory Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate Bevacizumab and Chemotherapy or Tarceva in Treating Recurrent or Refractory NSCLC (Non-Small Cell Lung Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: OSI2950g; NCT00098410 (obsolete NCT alias)
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Non-Small-Cell Lung Carcinoma; Neoplasm Recurrence, Local
Keywords: Recurrent or refractory non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Recurrence, Local; Recurrence | interventions — Bevacizumab; Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Avastin (bevacizumab)
Drug: Tarceva (erlotinib HCl)

SUMMARY:
This Phase II, multicenter, randomized trial is designed to make preliminary evaluations of the efficacy of combining bevacizumab with chemotherapy (docetaxel or pemetrexed) or Tarceva relative to chemotherapy (docetaxel or pemetrexed) alone in patients with previously treated advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically proven Stage IIIb with pleural effusion, or Stage IV, recurrent non-squamous NSCLC that is recurrent and unresectable
* Progression after one line of platinum-based chemotherapy (patients who have received prior docetaxel treatment are eligible to participate if there are no contraindications for pemetrexed treatment)
* Progression after previous adjuvant chemotherapy, if therapy was completed >= 6 months prior to randomization and the patient has received one line of therapy for recurrent disease
* (Optional) Availability of archival diagnostic tissue (paraffin tissue block or 2-10 unstained slides representative of the patient's primary cancer)
* ECOG performance status of 0, 1, or 2
* Life expectancy >= 3 months
* Measurable disease in accordance with RECIST
* Age >= 18 years
* Use of an acceptable means of contraception (potentially fertile men and women) or documentation of infertility

Exclusion Criteria:

* More than 30 days of prior treatment with an investigational or marketed agent that acts by EGFR inhibition (those with 30 or fewer days on an EGFR inhibitor without disease progression are eligible for enrollment)
* Treatment with an investigational or marketed agent that acts by anti-angiogenic mechanisms
* Previous treatment with more than one platinum-based chemotherapy
* Chemotherapy or radiotherapy within 28 days prior to randomization
* History of hemoptysis (> 1 teaspoon) or presence of a cavitary lesion
* Clinical history of Grade > 2 hematemesis within 6 months or Grade 1 hematemesis within 28 days prior to randomization
* History of serious systemic disease, including myocardial infarction within the last 6 months, uncontrolled hypertension (blood pressure > 150/100 mmHg on medication), unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or Grade II or greater peripheral vascular disease
* History or clinical evidence of CNS or brain metastases or CNS bleeding
* History or clinical evidence of hemorrhagic or thrombotic stroke within the 6 months prior to randomization
* Centrally located lesions and lesions that abut major blood vessels
* Ongoing treatment with full-dose warfarin (or its equivalent) or heparin (or its equivalent; e.g., Lovenox(R))
* In-patient surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization
* Minor surgical procedure, fine needle aspirations, or core biopsy within 7 days prior to randomization
* Anticipation of need for a major surgical procedure during the course of the study
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to take oral medication or requirement for IV alimentation or total parenteral nutrition with lipids, or prior surgical procedures affecting absorption
* Any of the following abnormal hematologic values (within 1 week prior to randomization): ANC <= 1,500 cells/uL; platelet count <= 100,000 cells/uL; Hemoglobin <= 9.0 g/dL; International normalized ratio (INR) > 1.5 x upper limit of normal (ULN)
* For patients who will receive docetaxel, any of the following abnormal liver function tests (within 1 week prior to randomization): Serum bilirubin greater than ULN; Albumin <= 2.5 g/dL; Serum ALT >= 1.5 x ULN; Serum AST >= 1.5 x ULN; Alkaline phosphatase >= 2.5 x ULN
* Other baseline laboratory values: Serum creatinine > 2.0 x ULN; Uncontrolled hypercalcemia ( > 11.5 mg/dL); Urinary protein/creatinine ratio >= 1 (spot urine) or clinically significant impairment of renal function; Estimated creatinine clearance < 45 mL/min (for patients who will receive pemetrexed)
* Any active systemic bacterial, fungal, or viral infection, including known hepatitis C and HIV
* Pregnant or breast-feeding
* Presence of another cancer within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix or non-melanomatous skin cancer
* Evidence of confusion or disorientation, or history of major psychiatric illness that may impair the patient's understanding of the Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2004-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and preliminary efficacy of combining bevacizumab with chemotherapy or Tarceva relative to chemotherapy alone on patients with previously treated advanced non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Vince O'Neill, M.D., Study Director — Genentech, Inc.
Locations (48):
- United States (48):
  - Comprehensive Blood and Cancer Center (TORI), Bakersfield, California
  - Bay Area Cancer Research Group, Concord, California
  - Virginia K. Crosson Cancer Center (TORI), Fullerton, California
  - California Cancer Center, Inc, Greenbrae, California
  - Wilshire Oncology Medical Group (TORI), Laverne, California
  - Pacific Shores Medical Group (TORI), Long Beach, California
  - UCLA Medical Center PVUB 3360, Los Angeles, California
  - Central Hematology Oncology Medical Group (TORI), Monterey Park, California
  - North Valley Hematology/Oncology Medical Group (TORI), Northridge, California
  - Ventura County Hematology-Oncology Specialists (TORI), Oxnard, California
  - Cancer Care Associates Medical Group (TORI), Redondo Beach, California
  - UC Davis Cancer Center, Sacramento, California
  - Kaiser Permanente/ San Diego, San Diego, California
  - Sansum Santa Barbara Medical Foundation Clinic (TORI), Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc (TORI), Santa Barbara, California
  - Kaiser Permanente Northern CA, Vallejo, California
  - San Diego Cancer Center Medical Group (TORI), Vista, California
  - Comprehensive Cancer Care Specialist at Boca Raton, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - The Florida Cancer Institute(TORI), Orlando, Florida
  - MD Anderson Cancer Ctr- Orlando, Orlando, Florida
  - Hematology and Oncology of Northeast Georgia, PC (TORI), Athens, Georgia
  - Medical Oncology Associates, PC (TORI), Augusta, Georgia
  - Suburban Hematology-Oncology Associates (TORI), Lawrenceville, Georgia
  - WellStar Cancer Research Office, Marietta, Georgia
  - Atlanta Cancer Care (TORI), Roswell, Georgia
  - Rush-Presbyteriam, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola Univ. Medical Center, Maywood, Illinois
  - Hematology Oncology Consultants, Naperville, Illinois
  - Oncoloy Hematology Associates of Central Illinois, PC (TORI), Peoria, Illinois
  - Norton Healthcare Louisville Oncology, Louisville, Kentucky
  - Ochsner Cancer Inst., New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Methodist Cancer Center-Oncology Research, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada (TORI), Las Vegas, Nevada
  - Summit Medical Group Overlook Oncology Center, Summit, New Jersey
  - Cancer Research of Long Island, Great Neck, New York
  - Northwestern Carolina Oncology and Hematology, Hickory, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Earle A. Chiles Research Institute, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Univ. of Pittsburgh Cancer Center Inst., Pittsburgh, Pennsylvania
  - University of Tenn. Cancer Ins, Memphis, Tennessee
  - The West Cancer Clinic, Memphis, Tennessee
  - M.D. Anderson, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Internal Medicine Associates of Yakima, Yakima, Washington